CLINICAL TRIAL: NCT01387373
Title: Intra-hepatic Chemotherapy With Oxaliplatin Every Second Week in Combination With Systemic Capecitabine in Patient With Non-resectable Liver Metastases From Breast Cancer. A Phase II Trial
Brief Title: Intra-hepatic Chemotherapy in Patient With Non-resectable Liver Metastases From Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dorte Nielsen (Other)
Responsible Party: Sponsor-Investigator, Dorte Nielsen, Responsible Party was entered in the old format as Dorte Nielsen, professor DMSci, Department of Oncology, Herlev Hospital., Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA 0919
Record Dates: First submitted 2011-05-31; First posted 2011-07-04 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Breast Cancer; Liver Metastases
Keywords: breast cancer; metastatic; liver metastases; intrahepatic; chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Oxaliplatin; Capecitabine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chemotherapy (Experimental)
  Interventions: Drug: oxaliplatin, capecitabine, trastuzumab

INTERVENTIONS:
Drug: oxaliplatin, capecitabine, trastuzumab — Oxaliplatin intrahepatic capecitabine + trastuzumab systemic
  Other Names: HAI

SUMMARY:
This is a phase II trial evaluating intra-hepatic chemotherapy with oxaliplatin every second week in combination with systemic capecitabine and in patients with a HER2-positive tumour in combination with trastuzumab (Herceptin®) in patient with non-resectable liver metastases from breast cancer.

Only patients without extrahepatic disease are included.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age > 18 years
* Performance status 0-1; expected survival ≥ 3 months
* Patient with histologically or cytologically confirmed locally advanced or metastatic adenocarcinoma of the breast
* Liver metastases not suitable for local treatment
* Extrahepatic disease should be excluded by PET-CT-scan.
* No progression on treatment with capecitabine.
* Prior treatment with taxane (adjuvant or for metastatic disease)
* Metastases < 70 % of the liver
* Neutrophile granulocytes > 1.5 x 109/l og thrombocytes > 100 x 109/l
* Bilirubin < 2.0 x UNL (upper normal limit).
* Creatinine-clearance > 30 ml/min.
* INR < 1.6.
* If the patient is HER2-positive:Baseline LVEF ≥ 50 %.

Exclusion Criteria:-

* History of chemotherapy within the 4-week period prior to the start of trial medication
* Other current or prior malignant disease except adequately treated and cured carcinoma in situ of the cervix or squamous cell carcinoma of the skin.
* Previous treatment with oxaliplatin
* Cytotoxic or experimental treatment within a 14 days period before start of trial medication
* The patient is not allowed to participate in other clinical trials.
* Any clinical symptoms suggesting peripheral neuropathy < or equal to grade 2 or CNS metastases (In case of clinical suspicion on CNS metastases a MR or CT scan should be performed within 4 weeks before inclusion
* Other severe medical conditions e.g. severe cardial disease or AMI < 1 year
* Presence of diseases which prevent oral therapy. • Patients with uncontrolled infection
* Pregnant or lactating women
* Women capable of childbearing not using a sufficient non-hormonal method of birth control
* Patients not able to understand the treatment or to collaborate.
* Prior serious or unsuspected reaction after treatment with fluoropyrimidine
* Known prior hypersensitivity reactions to the agents.

If the patient is HER2-positive:

• Dyspnoea in due to complication related to malignant disease e.g.lung metastases with lymphangitis or other conditions with need of supportive oxygen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-04; Primary Completion 2017-05-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 months after inclusion of last patient
  Number of patients with complete or partial response in the liver (RECIST version 1.1)Only patients with measurable disease are included in the protocol. Response rate number of patients with CR + PR divided with total number

SECONDARY OUTCOMES:
Time to progression a) Intrahepatic progression b) Extrahepatic progression | 6 months after inclusion of last patient
  Time from treatment start to progression of disease or death of any cause.
Number of patients suitable for local therapy (radiofrequency) | 6 months after inclusion of last patient
  Total number of patients receiving RF treatment or surgical treatment
Survival | 6 months after inclusion of last patient
  All patients in intent-to-treat population , calculated from start of treatment to death of any cause
Toxicity | 28 days after last patient last dose
  All patients who received at least one dose of study drug are evaluable for toxicity. CTC version 3.0 will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Nielsen, Professor, Principal Investigator — professor
Locations (1):
- Herlev Hospital, Herlev, Denmark